CLINICAL TRIAL: NCT06765993
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II/III Clinical Study of Isosorbide Oral Solution in the Treatment of Meniere's Disease
Brief Title: Efficacy and Safety of Isosorbide Oral Solution in Patients With Meniere's Disease
Acronym: MD
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lunan Better Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-YSLC-001
Record Dates: First submitted 2024-12-23; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Meniere´s Disease
Keywords: Meniere´s disease; Attack; Hearing loss; Tinnitus; Isosorbide
MeSH Terms: conditions — Hearing Loss; Tinnitus | interventions — Isosorbide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: Isosorbide oral solution
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isosorbide oral solution — 30 mL, TID
  Arms: Experimental group
Drug: Placebo — 30 mL, TID
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of isosorbide oral solution compared with placebo in people with unilateral Meniere's disease. A total of approximately 234 subjects will be enrolled in this study: 72 subjects in phase Ⅱ and approximately 162 subjects in phase Ⅲ. Patients were randomly assigned to either the experimental group or the control group. The randomization ratios for phase Ⅱ and phase Ⅲ were 1:1 and 2:1, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 and ≤65 years old.
2. Patients with unilateral Meniere's disease who meet the diagnostic criteria for Meniere's disease in the Guidelines for the Diagnosis and Treatment of Meniere's Disease (2017).
3. At least 3 episodes of vertigo caused by Meniere's disease within 6 months before enrollment.
4. Those who understand and voluntarily sign the informed consent.

Exclusion Criteria:

1. Patients who have had previous ear surgery for Meniere's disease.
2. People who suffer from vertigo caused by organic lesions of the external, middle or inner ear.
3. Patients with diseases that the investigators believe may limit the subjects' participation in this trial:

   * patients with acute intracranial hematoma;
   * patients with hypokalemia (serum potassium < lower limit of normal) or severe dehydration (needing infusion, or hospitalization, or life-threatening, requiring emergency treatment);
   * patients with acute pulmonary edema;
   * patients with hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure <60 mmHg during the screening period);
   * patients with severe cardiovascular and cerebrovascular diseases: such as New York Heart Association grade III or IV heart failure, myocardial infarction or unstable angina pectoris within the last 6 months, severe heart failure, progressive multifocal leukoencephalopathy, hypertension that is difficult to control with drugs (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥100 mmHg), etc.;
   * patients with major diseases of other important organs that affect their participation in this study.
4. Patients who need to use diuretics other than trial drugs for a long time after enrollment.
5. Patients with any of the following conditions are known or found in laboratory tests:

   * serum creatinine (Cr) level is not within the normal range;
   * human immunodeficiency virus (HIV) test is positive or has acquired immunodeficiency syndrome (AIDS);
   * active syphilis infection (positive Treponema pallidum antibody and positive non-specific syphilis antibody);
   * active hepatitis, hepatitis B: HBsAg and/or HBcAb are positive and HBV-DNA > 500 IU/mL or the lower limit of detection of the research center [only when the lower limit of detection of the research center is higher than 500 IU/mL]; hepatitis C: HCV antibody is positive and HCV-RNA is positive or greater than the upper limit of normal value.
6. Patients with known or suspected history of allergy to the investigational drug (isosorbide) and its excipients (sorbitol, lactic acid, saccharin sodium, propylparaben, butylparaben, orange flavor).
7. Those with a history of drug abuse or alcoholism within 6 months before enrollment.
8. Patients who have taken any prohibited drugs specified in this protocol for more than 1 week within 4 weeks before the first administration, including but not limited to vestibular suppressants (including antihistamines - promethazine, diphenhydramine, chlorpheniramine, etc., benzodiazepines - diazepam, lorazepam, clonazepam, etc., anticholinergics - scopolamine, atropine, glycopyrrolate, etc., and antidopamines - prochlorperazine, droperidol, etc.), betahistine, diuretics (including thiazide diuretics - hydrochlorothiazide, chlorthalidone, indapamide, indapamide sustained-release tablets, etc., loop diuretics - furosemide, torsemide, etc., potassium-sparing diuretics - amiloride, triamterene, etc.), glucocorticoids (including prednisone, methylprednisolone, betamethasone, beclomethasone propionate, prednisolone, hydrocortisone, dexamethasone, etc.).
9. Those who received intratympanic injection of gentamicin within the last year.
10. Patients who have received any other clinical trial drugs/devices within 30 days before the first dose.
11. Pregnant or lactating women, female patients or male patients' partners who plan to become pregnant during the study period and within 6 months after the last dose, and those who are unwilling to use a medically recognized effective contraceptive method (such as intrauterine contraceptive device or condom) during the trial.
12. Those who are judged by the researchers to be unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The changes from baseline in the number of vertigo attacks due to Meniere's disease during the treatment period | 3 months

SECONDARY OUTCOMES:
The changes in the number of vertigo attacks caused by Meniere's disease compared with the baseline at 6 months after the first administration. | 6 months after the first administration
The changes in the number of vertigo attacks caused by Meniere's disease compared with the baseline at 4-6 months after the first administration. | 4-6 months after the first administration
The changes in hearing from baseline 6 months after the first dose. | 6 months after first dose
  The assessment was made by subtracting the average hearing threshold of the worst pure tone audiometry test in the 6 months before treatment from the average hearing threshold of the worst pure tone audiometry test in the period 1 to 6 months after the first administration of the drug.
Patient-reported outcomes (PRO) during the treatment period were assessed using the Dizziness Handicap Inventory (DHI). | 3 months after the first dose
Patient-reported outcomes (PRO) during the treatment period were assessed using the Tinnitus Handicap Inventory (THI). | 3 months after the first dose
Patient-reported outcomes (PRO) were assessed using the Dizziness Handicap Inventory (DHI) at 6 months after the first dose. | 6 months after the first dose
Patient-reported outcomes (PRO) were assessed using the Tinnitus Handicap Inventory (THI) at 6 months after the first dose. | 6 months after the first dose

OTHER OUTCOMES:
The incidence and level of adverse events (AEs), serious adverse events (SAEs), abnormal laboratory test indicators, etc. | From the first dose to 30 days after the last dose
Change in tinnitus severity from baseline at 6 months after first dosing. | 6 months after the first dose
The change from baseline in the number of attacks due to Meniere's disease at 12 months after the first dose. | at 12 months after the first administration
The change in hearing compared to baseline at 12 months after first dose. | at 12 months after the first administration
  The assessment was made by subtracting the average hearing threshold of the worst pure tone audiometry test in the 6 months before treatment from the average hearing threshold of the worst pure tone audiometry test in the period 7 to 12 months after the first administration of the drug.
Patient-reported outcomes (PRO) were assessed using the Dizziness Handicap Inventory (DHI) at 12 months after the first dose. | at 12 months after the first dose
Patient-reported outcomes (PRO) were assessed using the Tinnitus Handicap Inventory (THI) at 12 months after the first dose. | at 12 months after the first dose
Changes in endolymphatic hydrops from baseline at 3 months after initial administration of isosorbide oral solution. | at 3 months after the first dose
Changes in endolymphatic hydrops from baseline at 6 months after initial administration of isosorbide oral solution. | at 6 months after first dose
  Only subjects who received maintenance dosing were evaluated.

IPD SHARING:
Plan to Share IPD: No
There are no plans to publish the findings in ICMJE journals.